CLINICAL TRIAL: NCT06652334
Title: Comparison of Spinal Anesthesia and Erector Spinae Plane Block in Terms of Pain Management, Perioperative Hemodynamic Changes, Morbidity and Mortality in Critically Adult Patients Undergoing Surgery Due to Femur Fracture
Brief Title: Comparison of Spinal Anesthesia and Erector Spinae Plane Block in Critically Adult Patients Undergoing Femur Surgery
Status: Completed | Type: Observational
Sponsor: Duzce University (Other)
Responsible Party: Principal Investigator, Özlem Ersoy Karka, Assistant Professor, Duzce University
Other Study IDs: drozlemersoy5
Record Dates: First submitted 2024-10-17; First posted 2024-10-22 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-06

CONDITIONS: Femoral Fractures
Keywords: Anesthesia, Spinal; Geriatric Anesthesia; Anesthesia and Analgesia; Nerve Block
MeSH Terms: conditions — Femoral Fractures; Agnosia | interventions — Anesthesia, Spinal

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Spinal anesthesia: 20 patients undergoing spinal anesthesia
  Interventions: Procedure: Spinal anesthesia
- Erector spinae plane block: 20 patients undergoing erector spinae plane block
  Interventions: Procedure: Erector spinae plane block

INTERVENTIONS:
Procedure: Spinal anesthesia — 20 patients undergoing spinal anesthesia
  Groups: Spinal anesthesia
Procedure: Erector spinae plane block — 20 patients undergoing erector spinae plane block
  Groups: Erector spinae plane block

SUMMARY:
The goal of this observational study is to compare the regional anesthetic methods (not including general anesthesia) -spinal anesthesia, erector spinae plane (ESP) block- which are in routine practice in critically ill adult patients operated for femur fracture, in terms of intraoperative and postoperative hemodynamics and clinical course, postoperative intensive care unit stay and hospitalization durations, pain scores, postoperative morbidity, and mortality.

Participants will undergo either spinal anesthesia or erector spinae plane block.

DETAILED DESCRIPTION:
Different anesthesia methods, including general and regional anesthesia, are used in operating rooms in daily practice. When general anesthesia is performed, the patient is rendered entirely unconscious by using intravenous and/or inhalation anesthetics, total sensory loss develops, and the patient's ventilation is provided by a mechanical ventilator. Regional anesthesia applications consist of blockage of nerve conduction by applying local anesthetics from different body parts without causing loss of consciousness. By using neuraxial anesthesia techniques - such as spinal anesthesia, epidural anesthesia, and caudal block - medulla spinalis-related neuronal blocking can be performed. Another regional anesthesia method whose use has expanded considerably in recent years is peripheral nerve blocks. This anesthesia method injects local anesthetic by targeting a specific plexus, nerve, or facia without any central nervous system blockage.

An essential part of intraoperative anesthesia management is planning analgesia for postoperative pain. It is aimed to provide analgesia with intravenous analgesics, central neuraxial blocks, or peripheral nerve blocks. Ensuring postoperative pain management has great importance in clinical practice because pain is associated with the patient's superficial breathing, prolonged immobilization, and noncompliant patients. Therefore, it is related to the development of atelectasis in the postoperative period and/or hypoxia-hypercarbia caused by inadequate gas exchange. In this situation where the patient cannot provide adequate respiration, the need for noninvasive mechanical ventilation may develop in the ward or intensive care unit where the patient is followed, closer clinical follow-up will be required, and the patient's hospitalization period will be prolonged. For this reason, it is one of the primary responsibilities to prefer anesthetic methods that help to provide optimal postoperative pain management.

Femoral fracture cases are primarily encountered in elderly patients with multiple comorbidities. Postoperative follow-up of these highly mortal fractures is often provided in intensive care units. In Turkish society, with an increasing elderly population, the long hospitalization periods of this patient group in the intensive care unit and their subsequent follow-up in the ward until they are discharged bring high healthcare costs. It has been shown in various studies in the literature that the anesthetic method is related to the length of hospitalization. Therefore, the clinical practices of anesthesiologists who frequently work with elderly patients in the operating room and intensive care are essential.

The clinician chooses the method of anesthesia, taking into account the type of operation, contraindications of the patient's clinical condition, pain management, postoperative follow-up conditions, and patient request. In critically ill patients with femoral fractures, the surgical procedure is successfully performed under general anesthesia, spinal anesthesia, or lumbar erector spinae plane (ESP) block. There are studies in which erector spinae plane (ESP) block applied from the lumbar region has been used as a primary anesthetic method that allows surgery in patients with femoral fractures.

In this study, the investigators aimed to compare the regional anesthetic methods (not including general anesthesia) -spinal anesthesia, erector spinae plane (ESP) block- which are in routine practice in critically ill adult patients operated for femur fracture in terms of intraoperative and postoperative hemodynamics and clinical course, postoperative intensive care unit stay and hospitalization durations, pain scores, postoperative morbidity, and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Agree to participate in the study
* Patients older than 65 years of age who are planning to undergo an operation for a femur fracture and who are in the ASA III and above risk group and for whom postoperative intensive care unit follow-up is foreseen
* Patients who agree to be operated under regional anesthesia

Exclusion Criteria:

* Patients who did not want to be included in the study
* Patients considered suitable for operation under general anesthesia
* Patients allergic to bupivacaine
* Patients with contraindications to neuraxial blockage (infection at the injection site, coagulopathy or other bleeding diathesis, severe hypovolemia, increased intracranial pressure, severe aortic stenosis, severe mitral stenosis)

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: After the patients who meet the specified criteria are informed about the study, 40 volunteers who agree to participate and sign an informed consent form will be included in the study.
  Volunteers will be randomized into 2 groups using a closed-envelope method. Group 1 will contain patients operated under spinal anesthesia, and Group 2 will contain patients operated under ESP block.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2024-10-20 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Pain scores | The VAS scores of the patients will be evaluated preoperatively, at 1 hour, 6 hours, 12 hours and 24 hours postoperatively.
  The Visual Analog Scale (VAS) is planned to be used for pain scoring. It will assess the severity of patients' pain in the preoperative and postoperative periods. It will be administered using a 10-centimeter line, with the words "no pain" on one side and "most severe pain" on the other.
  Patients will be asked to place a mark along the line at a level representing the intensity of their pain, which will then be measured in cm.
  The mark at 0 cm means "no pain," and the mark at 10 cm represents "the most severe pain the patient has ever sensed." Higher VAS scores mean the worst outcome.
  The patients' VAS scores will be evaluated preoperatively, at 1 hour, 6 hours, 12 hours, and 24 hours postoperatively.
Intraoperative sedation | The total dose of sedatives used along the operation will be calculated one time immediately at the end of the operation
  The total dose of sedatives used along the operation to maintain a BIS value between 80-90.
Intensive care unit length of stay | Through study completion, an average of 24 months.The intensive care unit length of stay will be calculated one time at the end of the intensive care unit stay, immediately at the timepoint of intensive care unit discharge.
  Time from end of the operation to discharge of the intensive care unit
Hospital length of stay | Through study completion, an average of 24 months.The ihospital length of stay will be calculated one time at the end of the hospital stay, immediately at the timepoint of the hospital discharge.
  Time from discharge of the intensive care unit to discharge of the hospital
Complications in the Intensive Care Unit | Complications will be recorded 1 time per day along the intensive care unit stay up to 90th day postoperatively.
  Clinical course - if any need for noninvasive/invasive mechanical ventilation, need for oxygen support, need for inotropes, development of acute kidney injury, state of consciousness, or additional complications- will be monitored and recorded at ICU (Intensive Care Unit).
Mortality | Mortality will be recorded 4 times up to 90th day postoperatively.: 1- at the time of discharge from the Intensive care unit, 2-at the time of discharge from the hospital 3- on the postoperative 30th day, 4- Mortality on the postoperative90th day
  In-hospital mortality, Intensive care mortality and Mortality after discharge. Patients will be followed up by telephone contact for mortality on the 30th and 90th postoperative days after discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Özlem Ersoy Karka, Ass. Prof., Study Director — Düzce University Faculty of Medicine
Locations (1):
- Duzce University Faculty of Medicine, Düzce, Düzce, Turkey (Türkiye)